CLINICAL TRIAL: NCT01059253
Title: Feasibility and Pilot Study of AdvanStep in Improving Balance in Elderly at Risk for Falls
Brief Title: Pilot Study of AdvanStep in Improving Balance in at Risk Elderly
Acronym: AdvanStep
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: equipment not functional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7170-HW-CTIL
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Impaired Balance in Elderly
Keywords: Falls; Balance; Elderly; Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training (Experimental): 15 training sessions
  Interventions: Other: AdvanStep training program - Turtle Pop

INTERVENTIONS:
Other: AdvanStep training program - Turtle Pop — Balance / mobility exercise program using the AdvanStep in a virtual reality context
  Other Names: AdvanStep Contoller p/n fg00002 rev. A1; Turtle Pop p/n gw00005 rev. A1

SUMMARY:
Elderly individuals are often at increased risks for falls. The AdvanStep is an interactive training exercise and balance device. The use of the AdvanStep will bring about a measurable improvement in the individuals balance in standardized measures.

DETAILED DESCRIPTION:
1. Feasibility study, assessing usability of the system and receiving feedback from the volunteers.
2. Structured treatment sessions twice per week after an initial assessment of balance and mobility on standardized tests.
3. Reassessment of balance and mobility after completion of 15 treatment sessions.
4. Treatment sessions will be supervised by physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80
* History of 2 falls in past 5 years, not requiring medical attention
* No acute orthopedic or neurological disorders
* No cognitive impairment affecting daily function.
* Adequate vision and hearing to see the computer screen and follow verbal commands.
* Unilateral stance test - inability to remain in unilateral stance for 25 seconds

Exclusion Criteria:

* Congestive heart failure or angina that limits physical activity
* Need for interventional medical treatment

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Performance on 4 square step test, Balance Evaluation Systems Test, 25 second unilateral stand test | On completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harold Weingarden, M.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel